CLINICAL TRIAL: NCT06280261
Title: The Struggle That Is Phenylketonuria : What Do The Patients and Caregivers Suffer From
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Dilara Demirel, MD, Hacettepe University
Other Study IDs: GO20/296
Record Dates: First submitted 2024-02-10; First posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Psychological Well-Being; Caregiver Burden; Life Stress
MeSH Terms: conditions — Psychological Well-Being; Caregiver Burden; Stress, Psychological | interventions — Psychological Tests

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: parenting stress index, Zarit burden scale, Rosenberg self esteem scale, stait trait anxiety inventory, struggles and difficulties questionnaire — Scales and questionnaires

SUMMARY:
Objective: To assess the stress levels and life hardships of phenylketonuria patients and their parents.

DETAILED DESCRIPTION:
Study Design: Between January 2020 - June 2020, a total of 156 phenylketonuria patients and their parents who arrived for their regular examinations were included. Parents were asked to fill the parenting stress index, Zarit burden scale and the strengths and difficulties questionnaire and children over the age of eleven were asked to fill the Rosenberg self-esteem scale, the stait-trait anxiety inventory and strengths and difficulties questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Phenylketonuria patients

Exclusion Criteria:

* BH4 metabolism disorde
* Other chronic illness
* Pregnancy

Ages: 6 Months to 35 Years | Sex: All
Age Groups: Child, Adult
Study Population: This study was carried out at Hacettepe University, İhsan Doğramacı Children's Hospital, Department of Metabolism, between January 2020 and June 2020. It was planned to include patients who were followed up with the diagnosis of phenylketonuria with diet or Sapropterin hydrochloride therapy, who didn't have BH4 metabolism disorder or any other health problem. Pregnant patients were also excluded
Sampling Method: Probability Sample
Enrollment: 156 (Actual)
Dates: Start 2020-05-27 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Rosenberg Self-Esteem Scale | 12 minutes
  Rosenberg Self-Esteem Scale was developed by Morris Rosenberg in 1960. It evaluates self-esteem and consists of 10 items in total. In the Likert-type scale, which includes positively and negatively charged items, 0-1 points are considered as high self-esteem, 2-4 points as medium self-esteem, and 5-6 points as low self-esteem.
Stait trait anxiety inventory | 45 minutes
  State-Trait Anxiety Inventory is an inventory that measures state and trait anxiety levels of children. It has been developed by Spielberges et. al in 1983. It consists of two questionnaires with a total of 40 questions, 20 that assesses the anxiety level stately, that is, how the child feels at that moment, and 20 that assesses how he feels constantly, that is, in general. The scale is in 3-point Likert type and is evaluated with 1-3 points according to symptom severityThe lowest score that can be obtained from the scales is 20, and the highest score is 60, higher scores indicate higher anxiety.
Strenghts and difficulties questionnaire | 30 minutes
  Strengths and Difficulties Questionnaire was developed by Goodman in 1997 to assess children's social, emotional and behavioral difficulties. There is a parent form for ages 4-17 and a child form for ages 11-17. It consists of 25 questions in total
Zarit burden scale | 25 minutes
  Zarit Burden Scale was developed by Zarit et al. in 1980. It is a 5-point Likert-type scale consisting of 22 questions that aims to measure the distress experienced by caregivers. Answers are scored between 0-4. A minimum of 0 and a maximum of 88 points can be obtained from the scale. The high score indicates the height of the distress experienced.
Parenting stress index | 20 minutes
  Parenting Stress Index aims to measure the stress experienced by parents in their relationships with their children. It is a 4-point Likert-type scale consisting of 16 questions in total. A minimum of 16 and a maximum of 64 points can be obtained from the scale. A high score from the scale indicates that parental stress is high.

CONTACTS AND LOCATIONS:
Overall Officials: Serap Sivri, Prof, Study Director — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Sihhiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-20): https://cdn.clinicaltrials.gov/large-docs/61/NCT06280261/Prot_SAP_000.pdf